CLINICAL TRIAL: NCT05168644
Title: Phase 1, Double-blind, Placebo-controlled, Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Safety and Pharmacokinetics Trial of Inhaled Niclosamide in Healthy Adult Subjects
Brief Title: Single Ascending Dose and Multiple Ascending Dose Study of Niclosamide Inhalation Powder in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TFF Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: TFF-N1-001
Record Dates: First submitted 2021-12-20; First posted 2021-12-23 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Part A: Eight (8) subjects will participate in each of the 3 dose escalations. Subjects will be randomized to receive either Niclosamide Inhalation Powder or placebo by inhalation (6 active, 2 placebo per group of 8).
  Part B: Eight (8) subjects will participate in each of the 2 dose escalations. Subjects will be randomized to receive either Niclosamide Inhalation Powder or placebo by inhalation (6 active, 2 placebo per group of 8).
Who Masked: Participant, Investigator
Masking Description: The investigators, study coordinators, study subjects and the Sponsor will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Drug: Niclosamide Inhalation Powder (Experimental): PART A (SAD): Niclosamide Inhalation Powder will be supplied as one to six capsules. Each capsule contains either 0.25 mg or 1 mg of Niclosamide Inhalation Powder and will be administered with a Plastiape RS00 Dry Powder inhaler. Doses may require multiple inhalations. All inhalations must be conducted within a 20-minute period.
  SAD subjects will receive a single dose of study medication. Subjects in Cohort 1 will receive 0.5 mg, Cohort 2: 2 mg, Cohort 3: 6 mg.
  PART B (MAD): Niclosamide Inhalation Powder will be supplied as one to six capsules. Each capsule contains either 0.25 mg or 1 mg of Niclosamide Inhalation Powder and will be administered with a Plastiape RS00 Dry Powder inhaler. Doses may require multiple inhalations. All inhalations must be conducted within a 20-minute period.
  MAD subjects will receive Niclosamide Inhalation Powder BID for a total of 9 doses. Subjects in Cohort 4 will receive 3 mg BID, Cohort 5: 6 mg BID.
  Interventions: Drug: Niclosamide Inhalation Powder
- Drug: Placebo (Placebo Comparator): PART A (SAD): Placebo will be supplied as one to six capsules. Each capsule contains Placebo inhalation powder and will be administered with a Plastiape RS00 Dry Powder inhaler. Doses may require multiple inhalations. All inhalations must be conducted within a 20-minute period.
  SAD subjects (Part A) will receive a single dose of Placebo.
  PART B (MAD): Placebo inhalation powder will be supplied as one to six capsules. Each capsule contains Placebo inhalation powder and will be administered with a Plastiape RS00 Dry Powder inhaler. Doses may require multiple inhalations. All inhalations must be conducted within a 20-minute period.
  MAD subjects (Part B) will receive Placebo inhalation powder BID for a total of 9 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Niclosamide Inhalation Powder — Investigational drug will be supplied as capsules, each capsule contains 0.25 mg or 1 mg of Niclosamide Inhalation Powder. The capsules will be administered with the provided breath actuated Plastiape RS00 Model 8 Dry Powder Inhaler device.
  Arms: Drug: Niclosamide Inhalation Powder
Drug: Placebo — Placebo will be supplied as capsules, each capsule will contain no active ingredient. The capsules will be administered with the provided breath actuated Plastiape RS00 Model 8 Dry Powder Inhaler device.
  Arms: Drug: Placebo

SUMMARY:
This is a Phase 1 (healthy adult volunteers), 2-part, double-blind, randomized, placebo controlled trial to evaluate the safety and pharmacokinetic (PK) profiles of escalating single doses of Niclosamide Inhalation Powder versus placebo (SAD part) and escalating multiple doses of Niclosamide Inhalation Powder versus placebo (MAD part). SAD part will be initiated first and includes a sentinel design. MAD part will not utilize a sentinel design unless the data monitoring committee requests the addition of sentinels. The MAD part will be initiated once the lowest doses from SAD part are deemed safe.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, 2 part double-blind, placebo-controlled trial to evaluate the safety and PK profiles of Niclosamide Inhalation Powder in a SAD/MAD study design.

Part A is a double-blinded, placebo-controlled, randomized, dose- ranging single dose study evaluating four different dose levels.

On Day 1 of each group, two selected subjects (sentinel subjects) will receive either Niclosamide Inhalation Powder or a matching placebo. Blood samples and safety measurements including Adverse Events (AEs) will be collected over 24 hour period following the drug administration. The safety results to be evaluated include AEs, concomitant medications, out of specification clinical laboratory results, vital signs, Electrocardiograms (ECGs), visual examinations, pulmonary function tests, pulse oximetry results and any new findings on physical examinations. If the administration is safe as deemed by Principal Investigator & Medical Monitor, the remaining six subjects will be dosed (5 dosed with Niclosamide Inhalation Powder and 1 dosed with matching placebo), with identical safety and PK procedures performed after minimum of 2 days interval. A minimum of 3 days will separate each dose escalation, with the remaining dose groups dosed in a sentinel fashion.

Part B is a double-blinded, placebo-controlled, randomized, dose- ranging multi-dose study evaluating two different dose levels. Dose level 1 of Part B can begin once the data monitoring committee reviews the safety data and indicates safety is present. Niclosamide Inhalation Powder will be administered twice daily (BID) × 9 doses. Blood samples for safety and PK will be collected throughout confinement, which is 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to use acceptable contraception or is not able to bear children.
2. Body mass index (BMI) within ≥ 18.0 kg/m2 and ≤ 30.0 kg/m2 at Screening (body weight of at least 50.0 kg and no more than120 kg at Screening).
3. Non-smoker or ex-smoker (stopped using nicotine products for at least 12 months prior to the first study drug administration and throughout the study).
4. Have no clinically significant diseases, including asthma, captured in the medical history or on the physical examination, visual examination, clinical laboratory assessments, and/or ECG.
5. A forced expiratory volume during the first second (FEV1) ≥ 80% at Screening and Check-in.

Exclusion Criteria

1. Female who is lactating, is pregnant or planning to become pregnant according to the pregnancy test at Screening or prior to the first study drug administration.
2. Is mentally or legally incapacitated or unable to provide informed consent.
3. History or presence of alcoholism or drug abuse within the past 2 years prior to the first study drug administration.
4. History or presence of hypersensitivity or idiosyncratic reaction to niclosamide or any portion of the placebo.
5. Has had surgery or any medical condition within 6 months prior to first study drug administration which may affect the absorption, distribution, metabolism, or elimination of the study drug, in the opinion of the PI or designee.
6. Use of albuterol or a similar bronchodilator.
7. Immunization with a COVID-19 vaccine in the 14 days prior to the first study drug administration.
8. Scheduled immunization with a COVID-19 vaccine (first or second dose) during the study that, in the opinion of an investigator, could potentially interfere with subject participation, subject safety, study results, or any other reason.
9. History or allergy of rare hereditary problems of galactose and/or lactose intolerance, lactase deficiency or glucose-galactose malabsorption.
10. Unable to refrain from or anticipates the use of:

    1. Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dosing and throughout the study.
    2. Seasonal use of albuterol or other similar inhalers throughout study participation, beginning 14 days prior to the first dosing or 5 half-lives, whichever is longer.
11. Use of St. John's wort in the 28 days prior to the first study drug administration.
12. Positive Screening results for tuberculosis, HIV Ag/Ab combo, hepatitis B surface antigen or hepatitis C virus tests, or a positive test for alcohol, cotinine, and/or drugs of abuse.
13. Participation in another clinical study within 30 days prior to the first study drug administration. The 30-day window will be derived from the date of the last study drug administration.
14. Had a treatment with another investigational drug within 5 times the elimination half-life, if known (eg, a marketed product) or within 30 days (if the elimination half-life is unknown) prior to the first study drug administration.
15. Donation of plasma in the 14 days prior to the first study drug administration.
16. Donation or loss of 500 mL or more of blood in the 56 days prior to the first study drug administration.
17. Demonstrates an inability to operate the inhalation device after training.
18. History or presence of any drug or food allergies.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-14 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Number of participants who experience Adverse Events (AEs), Serious Adverse Events (SAEs) and withdrawals due to AEs | Baseline through study completion, up to 43 days
  Number of AEs, SAEs, and discontinuation due to AEs
Number of participants who experience vital sign abnormalities | Baseline through study completion, up to 43 days
  Number of participants with potentially clinically significant vital sign values
Number of participants who experience pulse oximetry abnormalities | Baseline through study completion, up to 43 days
  Number of participants with potentially clinically significant pulse oximetry values
Mean change from baseline in forced expiratory volume (FEV1) | Baseline through study completion, up to 43 days
  Spirometry used to measure FEV1 lung function
Mean change from baseline in forced vital capacity (FVC) | Baseline through study completion, up to 43 days
  Spirometry used to measure FVC lung function
Mean change from baseline in FEV1/FVC ratio | Baseline through study completion, up to 43 days
  Spirometry used to measure FEV1 and FVC lung function
Mean change from baseline in QTcF changes via ECG | Baseline through study completion, up to 43 days
  Number of participants with potentially clinically significant ECG values
Number of participants who experience physical examination abnormalities | Baseline through study completion, up to 43 days
  Number of participants with potentially clinically significant physical examination findings
Number of participants who experience laboratory test abnormalities | Baseline through study completion, up to 43 days
  Number of participants with potentially clinically significant laboratory test results

SECONDARY OUTCOMES:
PK of Niclosamide in plasma: Area under the plasma-concentration time curve (AUC) | Baseline through study completion, up to 43 days
  Blood samples will be collected for plasma analysis
PK of Niclosamide in plasma: Area under the concentration time curve, from time 0 to the last observed non-zero concentration (AUC0-tlast) | Baseline through study completion, up to 43 days
  Blood samples will be collected for analysis
PK of Niclosamide in plasma: Maximum observed concentration (Cmax) | Baseline through study completion, up to 43 days
  Blood samples will be collected for analysis
PK of Niclosamide in plasma: Trough or minimum concentration (Ctrough) | Baseline through study completion, up to 43 days
  Blood samples will be collected for analysis
PK of Niclosamide in plasma: Concentration at the end of the dosing interval (Ct) | Baseline through study completion, up to 43 days
  Blood samples will be collected for analysis
PK of Niclosamide in plasma: Time to maximal observed concentration (tmax) | Baseline through study completion, up to 43 days
  Blood samples will be collected for analysis
PK of Niclosamide in plasma: Accumulation ratio (comparing Day 5 Cmax to Day 1 Cmax) | Baseline through study completion, up to 43 days
  Blood samples will be collected for analysis
PK of Niclosamide in plasma: Accumulation ratio (comparing Day 5 AUCtau to Day 1 AUC0-12) | Baseline through study completion, up to 43 days
  Blood samples will be collected for analysis
PK of Niclosamide in plasma: Area under the plasma-concentration time curve over the first 12 hours after dosing (AUC0-12) | Baseline through study completion, up to 43 days
  Blood samples will be collected for analysis
PK of Niclosamide in plasma: Area under the concentration time curve from time 0 extrapolated to infinity (AUC∞) | Baseline through study completion, up to 43 days
  Blood samples will be collected for analysis
PK of Niclosamide in plasma: Termination elimination half-life (t½) | Baseline through study completion, up to 43 days
  Blood samples will be collected for analysis
PK of Niclosamide in plasma: Apparent total body clearance (CL/F) | Baseline through study completion, up to 43 days
  Blood samples will be collected for analysis
PK of Niclosamide in plasma: Apparent volume of distribution during the terminal elimination phase (Vz/F) | Baseline through study completion, up to 43 days
  Blood samples will be collected for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Dale Christensen, PhD, Study Director — TFF Pharmaceuticals
Locations (1):
- Altasciences, Mount Royal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No